CLINICAL TRIAL: NCT05072470
Title: Benefits of an Assistive Listening Device for Speech Intelligibility in Noise
Brief Title: Benefits of Assistive Listening Device for Speech Intelligibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Hearts for Hearing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRF-70
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2021-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): Participants with bilateral moderate to severe sensorineural hearing loss
  Interventions: Device: Roger microphone; Device: Phonak Audeo hearing aid

INTERVENTIONS:
Device: Roger microphone — Commercially available transmitter microphone which sends distant speech signals to a receiver that is attached/embedded into hearing aids.
Device: Phonak Audeo hearing aid — Commercially available receiver-in-canal hearing aid

SUMMARY:
Speech intelligibility in noise will be evaluated in adults with moderate to moderate-severe sensorineural hearing loss, using an assistive listening device and hearing aid, and compared to speech intelligibility in noise using hearing aids alone.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18 or older with bilateral moderate to moderate severe sensorineural hearing loss, pure tone average must be between 40 and 69 dB HL (decibel Hearing Level)
* experienced hearing aid users
* symmetric hearing loss (no more than 15 dB difference between the ears at three contiguous frequencies)
* good written and spoken English language skills
* healthy outer ear as confirmed by otoscopy

Exclusion Criteria:

* contradictions to medical device noted upon otoscopy
* known hypersensitivity or allergy to materials of investigational device or comparator
* inability to produce reliable test results
* known psychological problems
* self reported symptoms of dizziness or vertigo

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hearts for Hearing, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 74 [48 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Bilateral Moderate to Severe Sensorineural Hearing Loss [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility in Noise
Description: The percent of correctly repeated words, when a list of 10 sentences is presented in noise. Ten sentences are presented at a certain loudness level while background noise is presented simultaneously at a specific loudness level. The number of words repeated correctly is calculated from the total number of words presented.
Time Frame: Day 1 of a one day study
Measure: Mean (Standard Deviation); unit: percentage of words correctly repeated
Arm/Group | Experimental
Number analyzed (Participants) | 10
percentage of words correctly repeated
  Percentage of words correctly repeated with hearing aid only at 0 dB SNR | 58 (26)
  Percentage of words correctly repeated with Roger system at 0 dB SNR | 80 (20)
  Percentage of words correctly repeated with hearing aid only at -5 dB SNR | 27 (17)
  Percentage of words correctly repeated with Roger system at -5 dB SNR | 50 (23)
  Percentage of words correctly repeated with hearing aid only at +5 dB SNR | 80 (22)
  Percentage of words correctly repeated with Roger system at +5 dB SNR | 87 (17)
Statistical Analysis 1: Comparison: Experimental; Speech intelligibility will be better with hearing aids plus Roger device, than with hearing aids alone when tested using standardized speech test at 0 dB SNR; Test type: Superiority — When p-value is adjusted for multiple comparisons, the level of statistical significance must be </= to .01666667 (.05/3); p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Experimental; Speech intelligibility will be better with hearing aids plus Roger device, than with hearing aids alone when tested using standardized speech test at -5 dB SNR; Test type: Superiority; p = .031, t-test, 2 sided — When p value is adjusted for multiple comparisons, the level of statistical significance must be </= to .01666667 (.05/3)
Statistical Analysis 3: Comparison: Experimental; Speech intelligibility will be equal or better with hearing aids plus Roger device than with hearing aids alone when tested using standardized speech test at +5 dB SNR; Test type: Superiority; p = .046, t-test, 2 sided — When p-values are adjusted for multiple comparisons, the level of statistical significance must be </= .01666667 (.05/3)

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT05072470/Prot_SAP_000.pdf